CLINICAL TRIAL: NCT02691104
Title: Use of the SMART COPD Physical Activity App in Pulmonary Rehabilitation: a Randomised Feasibility Study
Brief Title: Use of the SMART COPD Physical Activity App in Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); National Institute for Health Research: CLAHRC YH (Unknown); The Rotherham NHS Foundation Trust (Unknown); Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STH19149
Record Dates: First submitted 2016-02-12; First posted 2016-02-25 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Use of the app and Fitbit alongside 5-7 week pulmonary rehabilitation programme (plus goal-setting help from physiotherapist), and then app and Fitbit plus intermittent contact with physiotherapist for 8 weeks after pulmonary rehabilitation
  NB Randomisation is being deployed to test the practicality / acceptability of randomising for a larger RCT. It is not being used to assess the efficacy of the intervention in the current study
  Interventions: Device: SMART COPD app to promote physical activity in COPD. Used in conjunction with a Fitbit Charge
- Control (Other): Attend 5-7 week pulmonary rehabilitation programme (usual care) and wear blinded Fitbit during pulmonary rehabilitation and for 8 weeks afterwards
  NB Randomisation is being deployed to test the practicality / acceptability of randomising for a larger RCT. It is not being used to assess the efficacy of the intervention in the current study
  Interventions: Device: Control

INTERVENTIONS:
Device: SMART COPD app to promote physical activity in COPD. Used in conjunction with a Fitbit Charge — An app which allows users to set physical activity goals, monitors progress towards those goals, and provides feedback to users. Several options for types of physical activity (daily walk, daily step count, and aerobic / strengthening exercises) which can be tailored to the individual user. Designed to be used in consultation with a physiotherapist initially, and then used independently by the individual with COPD. The app will first be used alongside pulmonary rehabilitation (PR), with physiotherapist advice on exercises and setting goals. After PR the individual with COPD will receive weekly contact from a physiotherapist for the first 4 weeks, and then no contact for the second 4 weeks
  Other Names: The app has been developed by the research team and is not commercially available. A Fitbit® Charge pedometer will be used
  Arms: Intervention
Device: Control — Participants will follow the (usual care) PR programme. They will be asked to wear a blinided (cannot see step count) Fitbit Charge during the time they are on PR and then for 8 weeks afterwards
  Other Names: A Fitbit® Charge pedometer will be used
  Arms: Control

SUMMARY:
The investigators are carrying out a feasibility study to explore whether an app for physical activity in Chronic Obstructive Pulmonary Disease (COPD) is acceptable to people with the condition and to healthcare professionals who help patients manage the condition.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a long term lung condition which causes breathlessness, tiredness, coughing and chest infections. People with the condition often find it difficult to carry out day to day activities and to live a normal life. In recent years people with COPD have been encouraged to self-manage their condition, for example by increasing their physical activity, which could help them to live their life to the full. Recent advances in technology have the potential to help people do this. The SMART COPD 'app' which is being used in this study has been developed, based on previous research and the views of people living with the condition, to help people with COPD increase their physical activity. Physical activity is known to be important in helping people with COPD to enjoy better health and to carry out activities. The current study will investigate whether or not the app could be used alongside existing health services, and whether or not people with COPD, as well as healthcare professionals, find the 'app' acceptable and easy to use.

The investigators are working with three Pulmonary Rehabilitation (PR) teams in South Yorkshire (from Sheffield, Rotherham and Doncaster). PR is an education and exercise programme for people with lung conditions, which aims to teach people the skills to help them self-manage their condition. The first part of this feasibility study will investigate how PR is currently being delivered, and whether there would be any scope to include the app during and after PR to help people increase (or at least maintain) their physical activity levels longer term. This will be done by observing PR sessions, looking at how PR is delivered and referrals to the service, and through interactive workshops with healthcare professionals who deliver PR. The second part of the project will involve 'trying out' the app with a small group of people with COPD who are attending PR, to investigate whether the app is easy to use, whether any changes are needed, and the best way to use the app in the future. In order to determine whether the app successfully helps people with COPD to increase their physical activity levels, the investigators will need to carry out a much larger study in the future which compares use of the app with not having the app. The current feasibility project will help with planning this much larger study.

ELIGIBILITY:
Inclusion Criteria:

* A formal diagnosis of COPD;
* Attending a Pulmonary Rehabilitation (PR) course in Sheffield, Rotherham or Doncaster;
* Reasonable understanding of written and verbal English.

Exclusion Criteria:

* Not formally diagnosed with COPD;
* Deemed unable to attend standard PR;
* A cognitive impairment which prevents an individual giving informed consent;
* Does not understand written and verbal English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Usability and Acceptability of the intervention, as measured using qualitative interviews with staff and patient participants | Two years
  Thematic analysis of interviews will be used to explore participants' views on the usability and acceptability of the intervention.
Usability and Acceptability of the intervention, as measured using the System Usability Scale (SUS) (questionnaire with Likert-style questions) | Two years
  The SUS will provide an overall usability score for the intervention which will be comparable to other interventions which have used this scale.
Usability and Acceptability of the intervention, as measured using data on patterns of use for the app and Fitbit which are automatically logged by these devices. | Two years
  Data on patterns of use of the devices will help us determine whether there are parts of the intervention which are not used, or how different parts of the system are used (e.g. goal-setting strategies).

SECONDARY OUTCOMES:
Feasibility of conducting an RCT, including which outcome measures are of most relevance to people with COPD and healthcare professionals, whether those outcome measures would be feasible to use, and how feasible / acceptable randomisation would be | Two years
  As part of the feasibility study we will investigate a number of outcome measure options for a future large scale RCT, including physical activity logged by the devices (e.g. number of steps, whether goals are reached etc). We will also investigate a number of scales / questionnaires which measure different concepts which are potentially of interest (e.g. St George's Respiratory Questionnaire for quality of life, Exercise Self-Regulatory Efficacy Scale, EuroQol 5 Dimensions questionnaire for cost effectiveness etc), and acceptability of different outcomes measures. Acceptability of randomisation will be assessed through thematic analysis qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hawley, Principal Investigator — University of Sheffield
Locations (3):
- United Kingdom (3):
  - Doncaster and Bassetlaw Hospitals NHS Foundation Trust, Doncaster
  - The Rotherham NHS Foundation Trust, Rotherham
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield